CLINICAL TRIAL: NCT03851510
Title: Determination of the Prevalence and Severity of Expiratory Flow Limitation in Chronic Obstructive Pulmonary Disease Patients
Status: Terminated | Type: Interventional
Why Stopped: Study discontinued due to shifted business priorities.
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VectorEFLScreening-2018-10242
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Noninvasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants are first getting screened with Resmon Pro they then will be screened with the Vector ventilator for EFL. Those that screen positive with EFL with the Vector ventilator will be treated with the vector device with a 20 minute titration protocol.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Resmon Pro (Active Comparator): COPD participants will be first screened for Expiratory Flow Limitation using the Resmon Pro.
  Interventions: Device: Resmon Pro
- Vector Ventilator (Experimental): COPD participants will be screened again for Expiratory Flow Limitation using the Vector device, participants with EFL will undergo 20 minute titration protocol for therapy.
  Interventions: Device: Vector ventilator

INTERVENTIONS:
Device: Vector ventilator — The Vector ventilator is intended to provide non-invasive ventilatory support to treat adult patients with Obstructive Sleep Apnea (OSA), or Respiratory Insufficiency with the primary cause being COPD. This device is not intended for life support. It may be used to screened for the presence and abolishment of expiratory flow limitation. It is intended to be used within the home, institution/hospital, and diagnostic laboratory environments. The vector ventilator will titrate and treat EFL using non-invasive ventilatory support.
  Arms: Vector Ventilator
Device: Resmon Pro — The Resmon Pro uses the forced oscillation technique (FOT) which is a noninvasive method to measure the mechanical properties of the lung and airways during tidal breathing. In addition to measuring total impedance (resistance and reactance), the Resmon Pro can measure expiratory flow limitation which is a key index of respiratory obstruction
  Arms: Resmon Pro

SUMMARY:
Expiratory Flow Limitation (EFL) occurs when the airways become compressed, which usually results when the pressure outside the airway exceeds the pressure inside the airway. EFL can be detected using the Forced Oscillation Technique (FOT), which has been incorporated into a new screening feature in the Philips Respironics BiPAP Ventilator overall platform (Vector Non-Invasive (NIV) device). In this study, the Vector device will be used in a cross-sectional non-randomized epidemiology study to assess the prevalence and severity of expiratory flow limitation in a community COPD population. The study will also investigate how the presence of EFL may correlate with other physiological biomarker endpoints in the COPD patient. Participants will include 100 male and females with a diagnosis of COPD between the ages of 40 and 80. During the one-visit study, participants will undergo an EFL screening using the Vector device. If EFL is not detected during the screening after 5 minutes, the participant will not continue. If EFL is detected by the device, the participant will continue to wear it while it measures the level of therapy that is needed to eliminate EFL. Twenty minutes of pressure therapy will then be provided and the final Expiratory Positive Airway Pressure (EPAP) that is determined to abolish the participants EFL will be recorded. Participant characteristics (e.g. health history, behaviors, anthropometric, vitals, etc.) will be also be collected via questionnaires, medical record review, and physical exam. Future benefits of the study will be to gain a better understanding of the Vector screening feature and the characteristics of patients who present with varying degrees of EFL severity.

DETAILED DESCRIPTION:
This will be a cross-sectional, non-randomized epidemiology study designed to assess the prevalence and severity of expiratory flow limitation in a community COPD population. In the study we will also investigate how the presence EFL may correlate to other physiological biomarker endpoints in the COPD patient.

Schedule of Events:

Study Visit

* Once the participant arrives, the study will be explained in full detail. If the participant agrees, he/she will be consented into the study and the participant will be given a copy of the informed consent.
* Once consent is obtained, and eligibility is confirmed the following study related procedures will be conducted:
* Demographics: gender, date of birth, ethnicity, race, level of education will be collected.
* Current Medications: all current medications will be collected.
* Medical History Assessment: information will be collected regarding historical spirometry data, COPD history and other relevant medical history including the diagnosis of Sleep disordered breathing and Oxygen therapy usage. Chest computerized tomography (CT) scans will be collected if they have not been done within the past two years. A new CT scan will not be required.
* Physical examination with anthropometric data (weight, height and temperature) collected and vital signs to include Heart Rate (HR),Blood Pressure (BP), Respiratory Rate (RR), and Oxygen Saturation (SPO2) maintained at least 88% on room air, and chest auscultation.
* Review of inclusion/exclusion to ensure participant is eligible to continue
* Administration of Study Questionnaires
* Mask Fitting: Participants will have up to two mask fittings in order to determine the best possible masks while using the Vector NIV device during the EFL screening and titration.
* Spirometry testing will be performed for participants who have not had a test in the previous 6 months Resmon Pro EFL Measurement
* Participants will be required to wear nose clips during the measurement
* Participants will also be required to hold their cheeks during the measurement to prevent any air leaks around their mouth.
* While seated, participants will be instructed to breathe normally into the device for at least 30 seconds or until at least 10 breaths were successfully accepted by the device
* Participants will be asked to repeat test while in the supine or semi-recumbent position.

Vector EFL Screening/Determination and EPAP Titration

* EFL Determination: The participant will be asked to breathe quietly into the Vector device using the selected mask for 5 minutes in the seated position, and then an additional 5 minutes while in supine or semi-recumbent position. This device has the capability of detecting EFL. If it is determined that the participant does not have EFL by the device screening indicator, the participant will not continue with the EPAP titration.
* EPAP Titration: if it is determined by the Vector NIV device that the participant has EFL, the Vector NIV device will be changed from screening mode to therapy mode to delivery BiPAP therapy with the following settings.

Vector Device Settings:

* Pressure Support 6 cmH2O
* Max Pressure 26 cmH2O
* EPAP Min / EPAP Max 4 / 20 cmH2O
* The participants will then breathe on the Vector NIV device in the supine position (preferred) or semi-recumbent if needed for approximately an additional 20 minutes. During the additional 20 minutes of breathing, the device will automatically increase the EPAP (and concurrently and proportionally the IPAP) until the EFL is abolished (or falls below the predetermined EFL threshold).
* While the automatic EPAP Titration is being performed, all participants' SpO2 will be monitored via finger pulse oximetry.
* Patient must stay awake during the EPAP Titration. If the patient falls asleep, they will be woken by study staff.
* The Final EPAP that is determined to abolish the participants EFL will be recorded
* Participants will complete an EFL Vector device post questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years of age; < 80 years of age
* Ability to provide consent
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)

Exclusion Criteria:

* Any major non COPD uncontrolled disease or condition, such as congestive heart failure, malignancy, liver or renal insufficiency (that requires current evaluation for liver or renal transplantation or dialysis), amyotrophic lateral sclerosis, or severe stroke, or other condition as deemed appropriate by investigator as determined by review of medical history and / or participant reported medical history

  * Suffering from a COPD exacerbation at the time of data collection or in the 30 days prior to data collection
  * Self-reported Pregnancy
  * Employee or family member that is affiliated with Philips Respironics
  * History of bullous emphysema
  * History of pneumothorax
  * Evidence of acute sinusitis or otitis media
  * Hypotension
  * Participants at risk for aspiration of gastric contents
  * Epistaxis
  * Participants in respiratory failure
  * Inability to maintain a patent airway or adequately clear secretions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants That Were Consented.: All participants that were consented. If eligible, participants were screened for EFL with Resmon Pro and Vector devices.
Period: Overall Study
Arm/Group | All Participants That Were Consented.
Started | 57
Completed | 54
Not Completed | 3
Not completed — Screen Fail | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Includes only participants that were eligible. Baseline data was not available for the screened fail subject.
Arm/Group | All Participants That Were Consented.
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Overall Prevalence of Expiratory Flow Limitation
Description: The overall prevalence of EFL will be determined. This is defined as the percentage of participants exhibiting a DeltaXRS value greater than or equal to 2.8 using the Vector EFL device while supine. For purposes of this trial, overall prevalence includes indeterminate EFL and EFL.
Time Frame: 1 day
Population: One participant screened fail and data was not collected for the two discontinued participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants That Were Consented.
Number analyzed (Participants) | 54
Participants | 25
Statistical Analysis 1: Comparison: All Participants That Were Consented; All participants that were consented, eligible, and completed the Vector EFL screening (supine); Test type: Other — 95% confidence of prevalence measure; prevalence = 46.3, 95% CI 2-sided [32.6 to 60.4]

2. Secondary Outcome: Correlation of Titrated Final EPAP to Participants' Forced Expiratory Volume in One Second (FEV1)
Description: Correlation of titrated final EPAP (EPAP that is determined to abolish EFL) to patients' Forced Expiratory Volume in one second (FEV1).
Time Frame: 1 day
Population: Participants that were consented, eligible, screened positive for EFL, completed the titration and had spirometry data available.
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | All Participants That Were Consented.
Number analyzed (Participants) | 16
Spearman rank correlation coefficient | -0.278

3. Secondary Outcome: Correlation of Titrated Final EPAP to Participants' Screening DeltaXrs Value
Description: Correlation of titrated final EPAP (EPAP that is determined to abolish EFL) to participants screening DeltaXrs value
Time Frame: 1 day
Population: Participants that were consented, eligible, screened positive for EFL, and completed the titration.
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | All Participants That Were Consented.
Number analyzed (Participants) | 16
Spearman rank correlation coefficient | -0.427

4. Secondary Outcome: Percent of Participants With EFL Per the Resmon Pro That Have Their EFL Abolished During the Vector Screening.
Description: Percent of participants with EFL per the Resmon Pro that have their EFL abolished during the Vector screening. This will be calculated by the number of participants screened positive for EFL with the Resmon Pro who screened negative for EFL with the Vector device.
Time Frame: 1 day
Population: 46 participants were consented, eligible and screened for EFL with the Resmon Pro and Vector devices. Of those N=46, N=19 screened positive with the ResMon Pro device. Of those N=19, N=8 screened negative with the Vector device, resulting in 8/19 (42.1%).
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants That Were Consented.
Number analyzed (Participants) | 46
Participants
  Participants screened positive with Resmon Pro: number analyzed (Participants) | 19
  Participants screened positive with Resmon Pro: Participants screened positive with Vector | 11
  Participants screened positive with Resmon Pro: Participants screened negative with Vector | 8
  Participants screened negative with Resmon Pro: number analyzed (Participants) | 27
  Participants screened negative with Resmon Pro: Participants screened positive with Vector | 6
  Participants screened negative with Resmon Pro: Participants screened negative with Vector | 21

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the course of the study and up to 72 hours post study visit will be collected.
Arm/Group | All Participants That Were Consented.
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 1/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants That Were Consented. (N=57)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03851510/Prot_SAP_000.pdf